CLINICAL TRIAL: NCT02192658
Title: Disability and HIV: an Appraisal of the Vulnerability of People With Disabilities to HIV Infection in Two Main Cities of Sub-Saharan Africa
Brief Title: Disability and HIV: Vulnerability of People With Disabilities to HIV Infection in Sub-Saharan Africa
Acronym: HandiVIH
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Handicap International (Other); Institut de Recherche pour le Developpement (Other Government); Institut de Formation et de Recherche Démographique (Unknown); Forum Camerounais de Psychologie (Unknown); Centre de Recherche Internationale pour la Santé de l'Université de Ouagadougou (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS 12302 - HandiVIH
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV; Reproductive Health; Disability

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- People with Disability (PWD) (N= 850): PWD will be identified thanks to the disability screening tool developped by the Washington Group (WG). This tool is based on the WHO International Classification of Functionning (ICF).
  A stratified cluster sampling in 2 steps will be used in both, Yaounde and Ouagadougou. Each city will be divided in enumeration areas (EAs). First step : EAs will be drawn randomly with probability proportional to their size in number of households. Second step: in each EA, 30 households will be randomly drawn and each person living in these households will be screened for disability with the WG tool, according to the inclusion and exclusion criteria.
- Non-Disabled People (control group) (N= 850): For each PWD, 1 non-disabled control person will be randomly chosen from the census list of the same enumeration area. Control will also be matched on age and sex.

SUMMARY:
According to the recent World Report on Disability, around 15% of the world population lives with a disability and 80% of people with disabilities (PWD) live in developing countries. More and more evidence show that PWD are more likely to be poor, vulnerable to physical and sexual violence, and to have less access to education. Therefore, PWD are likely to have an increased risk for HIV infection, potentially being a key population in regard to this epidemic.

The vulnerability of PWD was recognized in 2007 by the United Nations Convention on the Rights of Persons with Disabilities. However, data on the extent how PWD are affected by HIV is still very limited. As a result, PWD are usually overlooked by National AIDS Control Programmes and few projects specifically targeting them have been developed.

Recognizing the need for appropriate and reliable data to help protect the rights of PWD and achieve a better inclusion of disability in National AIDS Control Programmes, the Institute of Research for Development (IRD), the Institut de Formation et Recherche Demographique (IFORD) and Handicap International (HI) propose this study that aims to provide quantitative and qualitative data on the vulnerability of PWD to HIV infection in Cameroon and Burkina Faso, in order to define if this vulnerable population is also a Key Population in relation to the HIV epidemic. This study adopts a multidisciplinary approach (quantitative and qualitative methods). Quantitative data are collected only in Cameroon.

Only the quantitative study is described here.

DETAILED DESCRIPTION:
OBJECTIVES:

The general objective of this study is to provide information on the vulnerability of PWD to HIV infection.

The objectives of the quantitative component of this study are:

Estimation of the HIV burden among PWD:

* To estimate the prevalence of HIV in PWD comprehensively and for each of the following disabilities 1) hearing 2) visual 3) mobility 4) cognitive (intellectual)
* To compare the HIV prevalence between PWD and non-disabled matched controls
* To assess the association between PWD's social network characteristics and the risk for HIV

Assessment of the knowledge, behaviour and practice toward HIV infection and sexual and reproductive health (including contraception) overall and for each of the impairment groups mentioned above:

* To describe and analyze the knowledge, attitude and behaviours related to HIV infection
* To compare the knowledge, attitude and behaviours between PWD and non-disabled matched controls
* To describe sexual and reproductive activities of PWD
* To describe and analyze the access and actual use of family planning methods in PWD

Access to HIV prevention and health careglobally and for each of the impairment groups mentioned above:

* To describe and analyze the determinants of and barriers to access to prevention and testing services
* To describe and analyze the determinants of and barriers to access to care
* To compare the access to services between PWD and non-disabled matched controls

Specific objectives related to disability:

* To describe the population of PWD in Yaoundé
* To describe and analyze the characteristics of the social networks of PWD

METHODOLOGY

Study design:

This is a cross sectionnal study assessing HIV prevalence, HIV risk factors and sexual & reproductive health of PWD compared to a control group of Non-Disabled People. PWD are sampled from the general population using a two-step sampling method. Eligible subjects are proposed an HIV test and to respond to a questionnaire on their Knowledge, Attitudes and Practices (KAP) in relation to HIV and SRH, on their social network and on their access to prevention and care services. The life-grid interview method is used to collect data on subject's history of social participation, employment, resources, sexual partnership and reproductive life. Controls are selected from the PWD's neighborhood.

Sample size:

850 disabled subjects and 850 non-disabled controls

Study location: Yaounde, Cameroon

Estimated planning or Study timetable :

Study start date: April 2014 (exploratory work) Total trial/study duration: 24 months

ELIGIBILITY:
For PWD:

Inclusion Criteria:

* Age 15 to 49 years
* WG criteria: ≥ 1 major impairment or 2 minor difficulties with an activity
* Informed consent given

Exclusion Criteria:

* Any severe disease that, according to the investigator, precludes the participation of the subject to ANY aspect of the study
* Temporary impairment (>1 year) which is likely to be cured quickly
* Subject consenting to none of the aspects of the study.

For Non-Disabled People (control group):

Inclusion criteria:

* Age 15 to 45 years in an interval of 5 years compared to the index PWD;
* Same sex as the index PWD;
* Not answering to the WG criteria for disability;
* Living in the same enumeration area as the Index PWD;
* Informed consent given.

Exclusion criteria:

* Any conditions, that - according to the interviewer - don't permit to participate at any part of the study;
* Subject consenting to none of the aspects of the study.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample:
  - PWD are identified thanks to the disability screening tool developped by the Washington Group (WG). This tool is based on the WHO International Classification of Functionning (ICF).
  A stratified cluster sampling in 2 steps is used in Yaounde. The city has been divided in enumeration areas (EAs). First step : EAs are drawn randomly with probability proportional to their size in number of households. Second step: in each EA, 30 households are randomly drawn and each person living in these households is screened for disability with the WG tool, according to the inclusion and exclusion criteria.
  - For each PWD, 1 non-disabled control person is randomly chosen from the census list of the same enumeration area. Controls are matched on age and sex.
Sampling Method: Probability Sample
Enrollment: 1610 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
HIV prevalence | 10 months
  HIV prevalence among People With Disability compared to Non-Disabled People. HIV serology will be assessed by rapid diagnostic tests.

SECONDARY OUTCOMES:
Risk factors | 10 months
  Risk factors to HIV and reproductive health behaviours among People with Disability compared to Non-Disabled People. Different risk factors (Knowledges - Attitudes - Practices) for HIV and reproductive health behaviours will be assessed in both groups, the people with disability group and the control non-disabled people group, through a questionnaire.

OTHER OUTCOMES:
Access to care | 10 months
  Access to services among People with Disability compared to Non-Disabled People. Access to reproductive health and HIV services will be assessed in both groups, through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DE BEAUDRAP, MD, PhD, Study Director — Institut de Recherche pour le Developpement (IRD); Gervais BENINGISSE, PhD, Study Director — Institut de Formation et Recherche Demographique (IFORD)
Locations (1):
- Yaoundé, Cameroon

REFERENCES:
- [Derived] De Beaudrap P, Pasquier E, Tchoumkeu A, Touko A, Essomba F, Brus A, Desgrees du Lou A, Aderemi TJ, Hanass-Hancock J, Eide AH, Mont D, Mac-Seing M, Beninguisse G. HandiVIH--A population-based survey to understand the vulnerability of people with disabilities to HIV and other sexual and reproductive health problems in Cameroon: protocol and methodological considerations. BMJ Open. 2016 Feb 4;6(2):e008934. doi: 10.1136/bmjopen-2015-008934. PMID 26846895